CLINICAL TRIAL: NCT07140185
Title: Evaluation of a Physical Activity Intervention on Sleep Quality, Mental and Physical Well-Being in Health Sciences Students: A Randomized Controlled Trial Comparing Regular Weekly Activity With a "Weekend Warrior" Pattern
Brief Title: Impact of a Physical Activity Intervention on Sleep Quality, Mental and Physical Well-Being in Health Sciences Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sfax (Other)
Responsible Party: Principal Investigator, Soumaya CHAABENE, Principal Investigator, University of Sfax
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMS110590-80-25
Record Dates: First submitted 2025-08-14; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sleep Quality; Sedentary Lifestlye; Physical Activity; Well-being
Keywords: Sedentary lifestyle; University students; Physical activity; Exercise intervention; Weekend Warrior; Sleep quality; well-being; Mental health; Fatigue; Randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity; Sedentary Behavior; Psychological Well-Being; Fatigue

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial uses a parallel-group design in which sedentary university students are randomly assigned to one of three groups: a regular weekly physical activity schedule group, a 'Weekend Warrior' physical activity group, or a control group. Each group participates concurrently throughout the 8-10 week intervention period. The parallel structure allows direct comparison of the effects of different physical activity patterns on sleep quality, mental well-being, and physical well-being.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Regular Weekly Physical Activity (Experimental): Participants in this group will engage in structured physical activity sessions three times per week, each lasting 50 minutes, over a period of 8 weeks. The sessions include a combination of aerobic exercises, supervised by trained instructors. The goal is to distribute the recommended weekly activity evenly across the week.
  Interventions: Behavioral: Regular Weekly Physical Activity Program
- Arm 2 - Weekend Warrior Physical Activity (Experimental): Participants in this group will perform the same total weekly physical activity as Arm 1, but concentrated in 2 sessions during the weekend. Each session lasts approximately 75 minutes and includes aerobic exercises, supervised by the same trained instructors.
  Interventions: Behavioral: Weekend Warrior Physical Activity Program
- Arm 3 - Control / No Intervention (No Intervention): Participants in this group will maintain their usual lifestyle without any structured physical activity intervention during the study period. After study completion, they may be offered the Regular Weekly physical activity program.

INTERVENTIONS:
Behavioral: Regular Weekly Physical Activity Program — Structured physical activity sessions three times per week, 50 minutes each, over 8 weeks. Includes aerobic exercises, supervised by trained instructors. Goal is to distribute the recommended weekly activity evenly.
  Arms: Arm 1 - Regular Weekly Physical Activity
Behavioral: Weekend Warrior Physical Activity Program — Same total weekly activity as Arm 1, but concentrated in 2 weekend sessions of 75 minutes each. Includes aerobic exercises, supervised by the same trained instructors.
  Arms: Arm 2 - Weekend Warrior Physical Activity

SUMMARY:
This randomized controlled trial aims to compare the effects of a regular weekly physical activity program versus a "Weekend Warrior" activity pattern on sleep quality, physical well-being, and mental well-being in sedentary university students. Participants will be randomly assigned to one of the intervention groups or to a control group and assessed at baseline and after the intervention.

DETAILED DESCRIPTION:
Sedentary behavior is a growing concern among university students and is associated with poor sleep quality, fatigue, and lower mental well-being. Physical activity interventions can improve these outcomes, but the optimal frequency and pattern of activity remain unclear. This randomized controlled trial will evaluate and compare the effects of a regular weekly physical activity schedule with those of a "Weekend Warrior" pattern, in which the recommended amount of exercise is concentrated in two sessions per week. Sedentary university students will be randomly assigned to one of two intervention groups or to a control group for an 8-10 week period. Sleep quality (measured by actigraphy), physical well-being, and mental well-being will be assessed before and after the intervention. The findings of this study may help to inform public health recommendations for physical activity patterns among young adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 25 years.
* Low level of physical activity, determined using the validated International Physical Activity Questionnaire (IPAQ) according to its scoring thresholds.
* Provided written informed consent.
* Available to participate in the entire intervention program and all planned assessments.

Exclusion Criteria:

* Current use of medications that may affect sleep quality or alertness (e.g., sedative hypnotics, sedative antidepressants, psychostimulants).
* History of serious medical conditions or any contraindication to moderate physical activity.
* Morbid obesity.
* Current pregnancy during the study period.
* Participation in another intervention program simultaneously.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency (Actigraphy) | Baseline (Week 0) and Post-intervention (Week 8)
  Sleep efficiency calculated as the ratio of total sleep time to time in bed, expressed as a percentage (%). ≥85% is considered good sleep, <85% indicates impaired sleep quality. Range: 0-100%. Higher percentages indicate better sleep efficiency.
Subjective Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline (Week 0) and End of Intervention (Week 8)
  Pittsburgh Sleep Quality Index total score ranges 0-21. Score ≤5 indicates good sleep quality, >5 indicates poor sleep quality. Higher scores indicate worse sleep.

SECONDARY OUTCOMES:
Psychological Well-Being (WHO-5 Well-Being Index) | Baseline (Week 0) and End of Intervention (Week 8)
  WHO-5 score ranges 0-25, converted to 0-100%. Higher scores indicate better well-being. Raw score <13 (<52%) suggests poor well-being.
Mental Health (Depression, Anxiety and Stress Scale, DASS-21) | Baseline (Week 0) and End of Intervention (Week 8)
  DASS-21 measures depression, anxiety, and stress. Each subscale score ranges 0-42; higher scores indicate greater severity.
Perceived Fatigue (Fatigue Severity Scale, FSS) | Baseline (Week 0) and End of Intervention (Week 8)
  FSS is a 9-item questionnaire. Items scored 1-7; final score = mean (range 1-7). Higher scores indicate more severe fatigue. Score ≥4 indicates clinically significant fatigue.
Functional Endurance (6-Minute Walk Test, 6MWT) | Baseline (Week 0) and End of Intervention (Week 8)
  6-Minute Walk Test measures distance (meters) walked in 6 minutes along a flat corridor. Higher distance indicates better functional endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Jihen JDIDI TRABELSI, Professor, Study Director — Faculty of Medicine of Sfax, Tunisia; Riadh DAHMEN, Professor, Study Director — Higher Institute of Sport and Physical Education of Sfax, TUNISIA
Locations (1):
- Private Faculty of Health Sciences Sfax, Tunisia, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
A decision on sharing individual participant data has not yet been made; plans will be determined after study completion and analysis.